CLINICAL TRIAL: NCT07130994
Title: Reduction or Elimination of Mitral Regurgitation With the SATURN Trans-septal TMVR System in Patients With Severe, Symptomatic Mitral Regurgitation (Cassini-US)
Brief Title: Reduction of Elimination of Mitral Regurgitation With the SATURN TMVR System (CASSINI-US)
Acronym: CASSINI-US
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InnovHeart (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0144
Record Dates: First submitted 2025-08-08; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Mitral Regurgitation; Heart Disease
Keywords: Transcatheter; Mitral Valve; Replacement
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Diseases

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- SATURN TMVR Cohort (Experimental)
  Interventions: Device: Mitral Valve Replacement

INTERVENTIONS:
Device: Mitral Valve Replacement — Implant of SATURN TS TMVR System for the treatment of moderate-severe or severe, symptomatic mitral regurgitation

SUMMARY:
CASSINI-US is a prospective, single-arm, multicenter early feasibility study enrolling up to 15 patients at up to 5 sites in the United States (US).

The purpose of the study is to evaluate the technical (implant) feasibility, and safety, and performance of the SATURN TS TMVR System for the treatment of moderate-severe or severe, symptomatic mitral regurgitation through a transcatheter approach.

Primary objectives evaluate the implant feasibility, and acute safety and performance of the SATURN TS TMVR System. The secondary objective and additional outcome measures characterize the long-term safety and performance of the SATURN TS TMVR System.

DETAILED DESCRIPTION:
The SATURN Bioprosthesis is designed to be implanted in the native mitral heart valve without open-heart surgery, extracorporeal circulation, cardiac arrest or removal of the failed native valve. The SATURN Bioprosthesis consists of the annular structure (Annular Segments) and the valve (SATURN Valve).

The valve supports a set of prosthetic leaflets that are the functional elements of the bioprosthesis. The valve is made of a self-expandable Nitinol frame supports three bovine pericardium leaflets. The valve is assembled with the annular structure through two connecting blocks mounted on the connecting arms of the stent.

The SATURN Delivery System and Accessories provides a transcatheter pathway to deliver the SATURN valve through the septum via the femoral vein. The SATURN Delivery System consists of an outer sheath, a guidewire delivery system, a valve delivery system and accessories.

The use of the SATURN TS System is carried out according to precise specifications and indications specified in the Instructions for Use (IFU) and is restricted to those physicians who have undergone dedicated training on use of the device.

Participants will be screened based on predefined inclusion and exclusion criteria. Eligible subjects will provide informed consent prior to any study-related procedures.

The clinical study designed to evaluate the safety, performance, and long-term clinical outcomes in adult patients with cardiac conditions. The study aims to collect comprehensive clinical data across patient population to support the understanding of procedural success, device-related outcomes, and patient recovery over time.

Participants will be followed from screening through five years post-procedure, with scheduled evaluations at the following timepoints: Screening, Baseline (pre-procedure), Intraprocedural, 24-48 hours post-procedure, 7 days or discharge, 1 month (±7 days), 3 months (±14 days), 6 months (±30 days), 1 year (±30 days), and annually through year five (±60 days).

Clinical assessments include physical examination, vital signs, and review of cardiac and antithrombotic medications. Functional status is evaluated using the Modified Rankin Scale, New York Heart Association (NYHA) classification, and the 6-Minute Walk Test. Quality of life is assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ). Risk stratification is performed at screening using EuroSCORE II and STS Risk Score.

Laboratory testing includes hematology, coagulation profiles, renal and liver function tests , and cardiac biomarkers such as NT-proBNP and plasma-free hemoglobin. Pregnancy testing is conducted at baseline for applicable participants.

Imaging and diagnostic testing includes transthoracic and transesophageal echocardiography (TTE/TEE), cardiac and vascular CT, gated cardiac CT at 6 months, 12-lead ECG, and intraprocedural assessments such as fluoroscopy, angiography, and right heart catheterization.

Safety endpoints include the incidence of adverse events (AEs), device deficiencies or malfunctions, and protocol deviations. The study is designed to generate robust clinical evidence supporting the intervention's safety, efficacy, and durability over time, and to inform future clinical practice and regulatory submissions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Symptomatic, moderate to severe or severe, functional or mixed, mitral regurgitation (≥ Grade 3+).
* NYHA functional Class ≥ II. If Class IV, patient must be ambulatory.
* Ability to tolerate oral anticoagulation.
* Ability to qualify for bailout surgery (which may include open heart surgery).
* High risk for open-heart mitral valve surgery due to age, co-morbidities or frailty, as determined by the Heart Team.
* Willing and able to complete study-related assessments and questionnaires.

Exclusion Criteria:

* Purely degenerative (organic/primary) (i.e. intrinsic valve lesions) mitral regurgitation.
* Excessive frailty or comorbid conditions that preclude the anticipated benefit of the mitral valve replacement.
* Life expectancy <1 yr. due to noncardiac conditions.
* Endocarditis in the 3 months prior to procedure date.
* Current admission with acute heart failure exacerbation.
* Dependency on inotropic agents or mechanical circulatory support.
* Untreated clinically significant CAD.
* Active systemic infection.
* Modified Rankin Scale ≥4 disability.
* Chronic renal failure defined as eGFR < 30 mL/min/m2 or on renal replacement therapy.
* Severe pulmonary arterial hypertension (PAH), defined as PASP > 70mmHg.
* Platelets < 90,000.
* COPD on home oxygen therapy deemed too high risk for intubation.
* Refuses blood transfusions.
* Documented bleeding or coagulation disorders (hypo- or hyper-coagulable states).
* Severe connective tissue disease under chronic immunosuppressive or cortisone therapy.
* Participating in other investigational studies likely to confound the results or affect the study.
* Unable or does not sign the study informed consent form.
* Patients classified as "vulnerable patients"

Cardiovascular Exclusion Criteria

* Myocardial infarction during prior 30 days.
* Stroke or TIA during prior 90 days.
* Severe extracardiac arteriopathy (safety measure for extra-circulatory support if surgical conversion is needed).
* Prior mitral valve treatment (e.g., valve repair or replacement, MitraClip, etc.), and/or anticipated mitral valve treatment prior to enrollment.
* Prior surgical mechanical valve AVR.
* Prior TAVI. -Need for any planned cardiovascular surgery or intervention (other than for MV disease) within 30 days post-index procedure.
* CRT, CRT-D, IPG or ICD implanted in previous 30 days.
* Cardiogenic shock, hemodynamic instability, Systolic Blood Pressure <90mmHg, Inotropic dependent or IABP/mechanical circulatory support.

CABG or PCI within previous 30 days.

* Inadequately treated for cardiac condition per applicable standards, such as for coronary artery disease, left ventricular dysfunction, mitral regurgitation, or heart failure, as reviewed by the Patient Screening Committee.
* Prior or planned heart transplantation (UNOS status 1).
* Physical evidence of right-sided CHF:

  1. Patients with ascites.
  2. Patients with anasarca (generalized edema / hydropsy).
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or other structural heart disease causing heart failure with the exception of dilated ischemic or non-ischemic cardiomyopathy.

Procedural Exclusion Criteria

* Known hypersensitivity or contraindication to procedural or post-procedural medication (e.g., contrast solution, anticoagulation therapy).
* Documented hypersensitivity to nickel or titanium.

Cardiac Imaging Exclusion Criteria (evaluated by Core Labs)

* Contraindications to TEE imaging
* Left ventricular EF ≤ 30% by echocardiogram.
* Severe mitral annular calcification, severe mitral stenosis, valvular vegetation or mass.
* Extensive mitral flail leaflets
* Evidence of new or untreated intracardiac thrombus, mass, or vegetation.
* Severe right ventricular dysfunction.
* Severe tricuspid regurgitation.
* Hemodynamically significant inter-atrial shunt (ASD).
* Severe aortic regurgitation or aortic stenosis.
* Anatomic ineligibility for SATURN Valve or SATURN TS procedure as determined by the Screening Committee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Technical (Implant) Success Endpoint | At completion of study procedure (Day 0)
  Presented as the n/N (%) of patients that meet the definition of Implant Success per protocol.
Freedom from Major Adverse Events Endpoint | 30 days from index procedure
  Freedom from (n/N, %) device-related or procedure-related major adverse events (MAE) which include:
  Cardiovascular death, Peri-procedural myocardial infarction, Disabling stroke, Major cardiac structural complication, Major vascular complication, and Mitral reintervention (operative or transcatheter) due to progressive or recurrent MR or device-related complications.
Mitral Valve Effectiveness Endpoint (reduction in MR grade) | 30 days post treatment
  Defined as the reduction of mitral regurgitation Grade to ≤1+ at 30 days.

SECONDARY OUTCOMES:
Mitral Valve Performance over time Endpoint | 5 years post index procedure
  Includes the following outcome measured at 30 days, 1 year and annually thereafter through 5 years post index procedure;
  -Reduction of MR grade compared to baseline and freedom from associated hemolysis

OTHER OUTCOMES:
Additional Safety Measurements (Incidence of AEs) | Measured at 30 days, 1 year and annually thereafter through 5 years post index procedure
  * All-cause mortality
  * All strokes
  * Acute kidney injury (AKI)
  * Mitral valve surgery or re-intervention
  * Re-hospitalizations for heart failure
Change in Quality of Life (KCCQ) | Baseline, 30 days, 3 months, 6 months, 1 year and annually thereafter through 5 years post index procedure
  The subject reported quality-of-life score (KCCQ) will be reported at each visit and compared to baseline. Scale 0-100, higher scores mean better outcomes.
Change in NYHA Classification | Baseline, 30 days, 3 months, 6 months, 1 year and annually thereafter through 5 years post index procedure
  The physician reported NYHA assessment (I-IV) will be reported at each visit and compared to baseline. Scale I-IV, higher score means a worse outcome.
Change in Six Minute Walk Test (6MWT) | Baseline, 30 days, 3 months, 6 months, 1 year and annually thereafter through 5 years post index procedure
  The distance walked (m) during the 6MWT will be reported at each visit and compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Torsten P Vahl, MD, Principal Investigator — Columbia University, New York, NY

IPD SHARING:
Plan to Share IPD: No